CLINICAL TRIAL: NCT05687591
Title: Left Atrial Appendage Occlusion With The Amplatzer Amulet Device: The Southeast Asia Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sarawak Heart Centre (Other)
Collaborators: InnoSignum (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Dr. Keng Tat Koh, Principal Investigator / Consultant Cardiologist and Electrophysiologist, Sarawak Heart Centre
Other Study IDs: Amulet-SEA-01
Record Dates: First submitted 2023-01-02; First posted 2023-01-18 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
Keywords: left atrial appendage occlusion; atrial fibrillation; Amplatzer Amulet
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients indicated for LAAO with the Amplatzer Amulet: All subjects who are indicated for LAAO with the Amplatzer Amulet are eligible for the study.
  Interventions: Device: Amplatzer Amulet Left Atrial Appendage Occlusion Device

INTERVENTIONS:
Device: Amplatzer Amulet Left Atrial Appendage Occlusion Device — The Amplatzer Amulet LAAO is a transcatheter, self-expanding device intended for use in preventing thrombus embolization from the left atrial appendage. The device is constucted from a nitinol mesh and consists of a lobe and a disc connected by a central waist. Polyester patches are sewn into both the lobe and disc to facilitate occlusion. The lobe has stabilizing wires to improve device placement and retention. The device has threaded screw attachments at each end for connection to the delivery and loading cables. The device has radiopaque markers at each end and at the stabilizing wires that permit visibility during fluoroscopy.

SUMMARY:
This is a prospective and retrospective, multicenter observational study where the study is being performed to explore on the short-term and long-term safety and efficacy of LAA occlusion with Amplatzer Amulet Device in Southeast Asia population on a real-world basis.

DETAILED DESCRIPTION:
The study is both retrospective and prospective, multicenter observational study for all patient indicated for LAAO with the Amplatzer Amulet device, involving subjects who had their occluder implanted, been recently implanted or intended to undergo the procedure may be considerd to participate in the study. The sample size is 100 and is based on the estimated number of recruitments from the participating centers. The study duration is 12 months of recruitment plus 1 year follow-up for outcomes. The outcomes are measured based on the objectives of the study:

Primary objective:

To explore on the short-term and long-term (1 year) safety and efficacy of LAA occlusion with the Amplatzer Amulet Device in Southeast Asia population on a real-world basis.

Secondary objective:

To compare the practice of LAA occlusion with Amplatzer Amulet Device in Southeast Asia population with the European registries.

Exploratory objective:

To explore the cost effectiveness of LAA occlusion with the Amplatzer Amulet Device in the Southeast Asia.

Descriptive statistics includes percentage, mean with standard deviation, or median with interquartile range will be reported, whichever appropriate. Categorical variables will be analysed using chi-square test or Fisher's exact test. Continuous variables will be analysed using independent (two variables only) or ANOVA test (more than two variables), or Mann-Whitney test (two variables only) or Kruskal-Wallis test (more than two variables) depending on the nature of underlying distributions. Time dependent outcome data will be analysed using Kaplan-Meier survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older
* Documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation
* At high risk of stroke or systemic embolism defined as CHA2DS2-VASc score of more than or equal to 3
* Deemed suitable for LAA occlusion by the treating physician, who might or might not be the investigator
* Able to comply with the required medication regimen post-device implant
* Able and willing to return for required follow-up visits and examinations

Exclusion Criteria:

* With active endocarditis or other infections producing bacteremia
* Where placement of the device would interfere with any intracardiac or intravascular structures
* Reversible cause of AF (i.e. secondary to thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
* Hypersensitivity to any portion of the device material or individual components of the Amulet LAA closure device
* Actively enrolled or plans to enroll in a concurrent clinical study in which the active treatment arm may confound the results of this trial
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the patient's ability to participate in the clinical trial or to comply with follow up requireemnts, or impact the scientific soundness of the clinical trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects who are indicated for LAAO with the Amplatzer Amulet are eligible for the study. Subjects who had their occluder implanted, been recently implanted or intended to undergo the procedure may be considerd to participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Device embolization | 1 year
  To determine if device embolization occurs (Yes/No). This is visualized through TOE or CT scan or TOE and CT scan
Device dislocation and device related thrombus | 1 year
  To determine if there is any device-associated thrombus occurs after the implantation of the occluder (Presence/Absence). This is visualized through TOE or CT scan or TOE and CT scan.
Peri-device leak | 1 year
  To determine if there is peri-device leak occurs after the implantation of the occluder (Yes/No). This is visualized through TOE or CT scan or TOE and CT scan.
Residual interatrial shunt | 1 year
  To determine if there is residual interatrial shunt occurs after the implantation of the occluder (Yes/No). This is visualized through TOE or CT scan or TOE and CT scan.
Mortality | 1 year
  To determine the mortality at 1 year after LAA occluder implantation
Ischemic Stroke and TIA | 1 year
  To determine the rate of ischemic stroke and TIA at 1 year after LAA occluder implantation
Major adverse bleeding event | 1 year
  To determine the rate of major adverse bleeding event at 1 year after LAA occluder implantation

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Keng Tat Koh, MBBS, Principal Investigator — Sarawak Heart Centre
Locations (1):
- Sarawak Heart Centre, Kuching, Sarawak, Malaysia

DOCUMENTS (2):
  • Study Protocol (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT05687591/Prot_000.pdf
  • Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT05687591/ICF_001.pdf